CLINICAL TRIAL: NCT00060151
Title: A Phase I, Open Label, Multiple Dose, Dose Escalation Study OF GW786034 In Patients With Solid Tumors
Brief Title: GW786034 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000299531; CASE-CWRU-100231; GSK-VEG10003; GSK-RM2002/00345/02; CWRU-GLAX-1Y02; CWRU-1Y02; CASE-100231
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2006-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Drug: pazopanib hydrochloride

SUMMARY:
RATIONALE: GW786034 may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth and by stopping blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of GW786034 in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of GW786034 in patients with advanced solid tumors.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the clinical response in patients treated with this drug.
* Evaluate the effect of this drug on biomarkers of angiogenesis activity in order to estimate activity and to determine the minimum biologically active dose in these patients.

OUTLINE: This is an open-label, nonrandomized, dose-escalation, multicenter study.

Patients receive oral GW786034 twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 2-6 patients receive escalating doses of GW786034 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 21 days.

PROJECTED ACCRUAL: Approximately 30-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor
* Refractory to standard therapy or for which no standard therapy exists
* No untreated leptomeningeal or brain metastases

  * Previously treated brain metastases are allowed if currently asymptomatic and patient is off steroids and antiseizure medications for more than 3 months before study entry

PATIENT CHARACTERISTICS:

Age

* 21 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2 times upper limit of normal (ULN) (5 times ULN if tumor involvement)

Renal

* Creatinine clearance at least 60 mL/min

Cardiovascular

* No uncontrolled hypertension (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg on 2 consecutive measurements separated by 1 week)
* No arterial or venous thrombosis (including cerebrovascular accident) within the past 3 months
* No myocardial infarction within the past 3 months
* No unstable angina within the past 3 months
* No cardiac angiopathy or stenting within the past 3 months
* No cardiac pacemaker

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 21 days after study treatment
* Able to swallow and retain oral medication
* Good venous access
* No prior or concurrent gastrointestinal disease
* No prior or concurrent condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug
* No other unstable, pre-existing major medical condition
* No orthopedic pins or rods or other embedded metal that would preclude undergoing an MRI
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy
* Concurrent epoetin alfa allowed
* No concurrent anticancer biologic therapy

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No concurrent anticancer cytotoxic chemotherapy

Endocrine therapy

* See Disease Characteristics
* More than 4 weeks since prior hormonal or steroid therapy (other than replacement)
* No concurrent anticancer hormonal therapy (except for replacement)
* No concurrent dexamethasone or prednisone

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No concurrent anticancer radiotherapy

Surgery

* More than 4 weeks since prior major surgery
* No concurrent surgery for cancer

Other

* Recovered from prior therapy
* More than 4 weeks since prior investigational agents
* More then 28 days since prior alteration of antihypertensive medications
* Concurrent bisphosphonates allowed
* No other concurrent anticancer therapy
* No concurrent antidepressants (e.g., amitriptyline, fluoxetine, or fluvoxamine)
* No concurrent oral hypoglycemics (e.g., glipizide, glyburide, rosiglitazone, or tolbutamide)
* No concurrent therapeutic anticoagulation (e.g., warfarin at therapeutic doses)

  * Low-dose anticoagulation for prophylaxis allowed
* No concurrent cyclosporine
* No concurrent grapefruit juice
* No concurrent amiodarone, mibefradil, phenobarbital, or pioglitazone
* No concurrent Hypericum perforatum (St. John's Wort)
* No concurrent rifabutin or diethyldithiocarbamate
* No concurrent gestodene, mifepristone, or modafinil
* No concurrent herbal supplements, vitamins, or non-traditional compounds

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-12; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity assessed weekly during treatment

SECONDARY OUTCOMES:
Disease response every 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Study Chair — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Result] Hurwitz HI, Dowlati A, Saini S, Savage S, Suttle AB, Gibson DM, Hodge JP, Merkle EM, Pandite L. Phase I trial of pazopanib in patients with advanced cancer. Clin Cancer Res. 2009 Jun 15;15(12):4220-7. doi: 10.1158/1078-0432.CCR-08-2740. Epub 2009 Jun 9. PMID 19509175